CLINICAL TRIAL: NCT01622998
Title: Self-directed Titrated Transdermal Nicotine Patch Versus Standard Treatment for Smoking Cessation in Smokers Motivated to Quit
Brief Title: Self-directed Titrated Transdermal Nicotine Patch Versus Standard Treatment for Smoking Cessation
Acronym: STEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA7025
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Smoking Cessation
Keywords: Pharmacotherapy; Titration; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard transdermal NRT group (UC) (Active Comparator): 10 week standard transdermal nicotine replacement therapy patch protocol
  Interventions: Drug: NicoDerm Patch
- Titrated transdermal NRT group (EXP) (Experimental): 10 week titrated transdermal nicotine replacement therapy patch dose regimen based on smoking history with the option to increase dose, if withdrawal symptoms are unmanageable.
  Interventions: Drug: NicoDerm Patch; Drug: Nicorette Inhaler

INTERVENTIONS:
Drug: NicoDerm Patch — Dosage: 21mg patch; 14mg patch; 7 mg patch Frequency: NRT patch application once per day Duration: 10 week treatment period
  *Titration for experimental group (NRT+) based on smoking history, and option to increase dose if withdrawal symptoms are unmanageable.
  Other Names: Nicoderm 21mg, NPN: #02093146; Nicoderm 14mg, NPN: #02093138; Nicoderm 7mg, NPN: #02093111
Drug: Nicorette Inhaler — Nicorette Inhaler: Box, 42 cartridges (4mg/cartridge) Dosage: Ad libitum Maximum dosage: 6-12 cartridges/day
  Other Names: Nicorette Inahler, NPN: #02241742
  Arms: Titrated transdermal NRT group (EXP)

SUMMARY:
The primary aim of this research study is to determine whether titrated, patient-directed transdermal patch NRT, based on smoking history and symptoms of nicotine withdrawal, improves long-term rates of smoking cessation in patients motivated to quit smoking when compared to patients using the standard transdermal NRT patch protocol. The following hypothesis will be tested: CO-validated continuous abstinence rate at 52 weeks post target quit date will be higher for the titrated, self-directed NRT group compared to the standard NRT treatment group.

DETAILED DESCRIPTION:
Participants will be recruited from the UOHI Smoking Cessation Clinic and via media advertisements. Following their baseline assessment, participants will be randomly assigned to one of two groups:

1. 10-week standard treatment of transdermal nicotine replacement therapy (NRT);or
2. 10-week titrated transdermal nicotine replacement therapy (NRT) treatment with additional NRT product (NRT+)

Participants assigned to the "NRT" standard treatment group will follow a 10-week regimen of nicotine patches alone.

Participants assigned to the "NRT+" titrated treatment group will follow a 10-week regimen of tailored patch dosage. Participants will also be provided with the Nicorette inhaler.

All participants will receive five 15-minute counselling sessions from a smoking cessation counsellor. These sessions occur at 1, 3, 5, 8 and 10 weeks post target quit date. Counselling sessions will focus on practical counselling (problem solving and skills training) and social support.

During the treatment phase, participants will complete questionnaires measuring withdrawal symptoms, self-efficacy, use of cessation resources and the Beck Depression Inventory (BDI-II) at weeks 1, 3, 5, 8 and 10. These questionnaires will also be completed at 26 and 52 weeks post target quit date.

ELIGIBILITY:
Inclusion Criteria:

1. Current smoker (≥ 10 cigarette per day);
2. 18 years of age or older;
3. Willing to set a date to quit smoking within the 30 days following the baseline assessment;
4. Participant is willing to return to the UOHI for follow-up examination;
5. Participant is willing to provide informed consent;
6. Motivated to quit smoking.

Exclusion Criteria:

1. Participant is unable to read and understand English or French;
2. Participant is pregnant, lactating or planning to become pregnant during the study period;
3. Participant has attempted to quit smoking in the previous month with the support of medication for >72 hours;
4. Participant is currently using a smoking cessation medication (e.g., NRT, Bupropion, Varenicline,Clonadine, Notriptyline);
5. Participant has contraindication(s) to nicotine replacement therapy (allergy to adhesive, life-threatening arrhythmias (e.g., tachycardia);
6. Participant is during the immediate post-myocardial infarction period (i.e. incident has occurred within the last 10 days);
7. Severe or worsening angina pectoris;
8. Subject has had a recent cerebral vascular accident (i.e. incident has occurred within the last 10 days);
9. Participant currently suffering with depression (BDI-II ≥20);
10. Participant who has been diagnosed with depression or treated with an antidepressant in the past 12 months;
11. Past or present history of psychosis (Schizophrenia, Schizophreniform or Delusional Disorders),panic disorder, or bipolar disorder;
12. Drug or alcohol abuse or dependence in the past year;
13. Member of the participant's household is already participating in the study or in the "Quit Smoking in the 'Real World'" study;
14. Participant is currently participating in or already receiving counseling or follow-up for smoking cessation.

13.) Participants who in the opinion of the investigator will be unlikely to commit to a year-long study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Validated continuous abstinence rate at week 52 | Week 52
  Self-reported continuous abstinence at week 52 post target quit date will be confirmed with a carbon monoxide breath test.

SECONDARY OUTCOMES:
Validated continuous abstinence rates at weeks 10 and 26 weeks and seven day point prevalence of abstinence rates at weeks 10, 26 & 52 | weeks 10, 26 and 52
  Self-reported continuous abstinence rates will be validated with a carbon monoxide breath test at weeks 10 and 26 post target quit date.
  Self-reported seven day point prevalence of abstinence will be validated at week 10, 26 and 52 weeks post target quite date.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pipe, CM, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Hughes JR, Keely J, Naud S. Shape of the relapse curve and long-term abstinence among untreated smokers. Addiction. 2004 Jan;99(1):29-38. doi: 10.1111/j.1360-0443.2004.00540.x. PMID 14678060
- [Background] Clinical Practice Guideline Treating Tobacco Use and Dependence 2008 Update Panel, Liaisons, and Staff. A clinical practice guideline for treating tobacco use and dependence: 2008 update. A U.S. Public Health Service report. Am J Prev Med. 2008 Aug;35(2):158-76. doi: 10.1016/j.amepre.2008.04.009. PMID 18617085
- [Background] Slovinec D'Angelo ME, Reid RD, Hotz S, Irvine J, Segal RJ, Blanchard CM, Pipe A. Is stress management training a useful addition to physician advice and nicotine replacement therapy during smoking cessation in women? Results of a randomized trial. Am J Health Promot. 2005 Nov-Dec;20(2):127-34. doi: 10.4278/0890-1171-20.2.127. PMID 16295704
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995